CLINICAL TRIAL: NCT06706050
Title: Clinical Evaluation of Lactobarriome 5% Cream's Efficacy on Dry Skin for Improving Skin Hydration and Transepidermal Water Loss, Relieving Pruritus, and Altering the Skin Microbiome
Brief Title: Clinical Therapeutic Potential of Novel Microbiome LP-51 on Xerosis Individual Based on Xerosis-microbiome Index
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ho-Yeon Song (Other)
Collaborators: National Research Foundation of Korea (Other); Ministry of Trade, Industry and Energy (Unknown); Soon Chun Hyang University (Other)
Responsible Party: Sponsor-Investigator, Ho-Yeon Song, Professor, Soon Chun Hyang University
Organization: Soon Chun Hyang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S23004-01
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Xerosis
Keywords: xerosis-microbiome index; Microbiome therapeutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: LP-51 (Experimental): test substance was applied on participants
  Interventions: Biological: Microbiome Therapeutic LP-51
- Arm 2: Placebo (Placebo Comparator): cream without active substance (M23004-03) was applied on the participants
  Interventions: Other: placebo cream (M23004-03)

INTERVENTIONS:
Biological: Microbiome Therapeutic LP-51 — Microbiome therapeutics LP-51 was applied on the individuals suffering from xerosis
  Arms: Arm 1: LP-51
Other: placebo cream (M23004-03) — placebo cream (M23004-03) was applied on the participants
  Arms: Arm 2: Placebo

SUMMARY:
The purpose of this clinical trial is to assess the skin hydration and transepidermal water loss improvement, pruritus relief, and microbiome alteration effects of a Lactobacillus sp. product (Lactobarriome 5% cream) compared to a placebo cream to prove the skin improvement effects of Lactobarriome 5%, which is a nature-friendly material derived from intravaginal microflora that can replace chemical components commonly used as ingredients for existing cosmetics.

The impact of Lactobarriome 5% cream, formulated with LP51 culture filtrate, on dry skin was assessed through a 4-week double-blind clinical trial. Participants were selected based on predefined inclusion and exclusion criteria. Using a simple randomization method, participants were assigned to either the experimental group (receiving the test formulation) or the control group (receiving a placebo). The products were applied twice daily-morning and evening-to a 3 cm area on both the proximal and distal sides of the designated arm's crook. Clinical evaluations were conducted at baseline, as well as after 2 weeks and 4 weeks of product use. These assessments included visual inspections, subjective pruritus evaluations, skin hydration levels, and transepidermal water loss (TEWL) measurements, all performed by a skincare professional. Furthermore, magnified images were captured using a Folliscope, and skin samples were collected to analyze microbial changes post-treatment. Before application, the designated arm was washed with water and allowed to rest for 30 minutes under controlled conditions (22±2°C, 50±10% relative humidity).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, including men and women, aged 19-70
* Without acute or chronic diseases (excluding atopic dermatitis)
* Individuals suffering from dry skin and itchiness in the test area (crook of the arm)
* Those with objectively proven skin barrier damage demonstrated by a transepidermal water loss (TEWL) value of ≥12 g/h/m² and a skin hydration value below 35 (Corneometer measurement)
* Individuals who provided voluntary informed consent
* Those who agreed to comply with study visits and observations

Exclusion Criteria:

* Individuals with active skin diseases requiring treatment
* Those with an ESIF score >6
* Individuals with a history of antibiotic, steroid, immunosuppressant, antihistamine, or retinoid use, or phototherapy within the last 4 weeks
* Individuals who used skin disease-related supplements or moisturizers within 2 weeks
* Those participating in other clinical trials within the last 4 weeks
* Individuals with frequent exposure to UV light
* Pregnant or lactating women
* Those planning pregnancy during the trial period
* Any other factors deemed unsuitable by the investigator

Ages: 21 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Improvement of skin hydration and transepidermal water loss, and relieving pruritus | From enrollment to the end of treatment at 4 weeks
  A 4-week double-blind clinical trial involving 43 participants suffering from xerosis was conducted to evaluate the therapeutic potential of Microbiome therapeutic LP51. To serve this purpose, Lactobarriome 5% cream containing LP51 culture filtrate was applied on the dry skin for 4-week. A random allocation chart (Simple Randomization method) was used to assign participants to the experimental group (test formulation) or control group (placebo).
  The volunteers applied the product twice daily (morning and evening) to a 3 cm area proximal and distal to the crook of the designated arm. Clinical parameters were evaluated at baseline, after 2 weeks, and after 4 weeks of use. Visual assessments, subjective pruritus evaluations, skin hydration measurements, and TEWL measurements were conducted at every visit by a skin professional. Additionally, magnified photographs were taken using a Folliscope, and skin samples were collected to assess microbial changes after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang University Probiotics Microbiome Convergence Center (PMC) Skin Clinical Evaluation Research Institute, Asan, Chungnumdo, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF